CLINICAL TRIAL: NCT05648760
Title: Simulation-based Training Improves Medical Student Competency in Communicating Bad News to Patients: A Randomized Controlled Trial
Brief Title: Simulation-based Training Improves Competency in Communicating Bad News
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jingyuan,Xu, Principal Investigator, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2022ZDYYLL01
Record Dates: First submitted 2022-12-05; First posted 2022-12-13 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Simulation of Physical Illness
Keywords: simulation; competency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual training (Other): Participants randomized to the control condition received a standard training of how to communicate bad news to patients
  Interventions: Behavioral: Simulation training
- Simulation training (Experimental): Participants randomized to the simulation training group received simulation training based on a standard training of how to communicate bad news to patients
  Interventions: Behavioral: Simulation training

INTERVENTIONS:
Behavioral: Simulation training — Participants randomized to the simulation condition received simulation training based on a standard training of how to communicate bad news to patients

SUMMARY:
Delivering bad news is a task that doctors encounter daily in most medical practices, especially in Intensive Care Unit, where morbidity and mortality are high. The objective of this project was to demonstrate effectiveness of an educational program using simulation-based training intervention to teach medical students to deliver bad news and communicate more effectively with families.

DETAILED DESCRIPTION:
Delivering bad news is a task that doctors encounter daily in most medical practices, especially in Intensive Care Unit, where morbidity and mortality are high. The term "bad news" refers to any information transmitted to patients or their families that directly or indirectly involves a negative change in their lives or view of their future. Existing reports show that practicing doctors and residents lack confidence and skill in performing this task, and most have never received any formal training. Breaking bad news is a complex task requiring many skills including communication, responding to emotional reactions, and involving the family members.

The objective of this project was to demonstrate effectiveness of an educational program using simulation-based training intervention to teach medical students to deliver bad news and communicate more effectively with families. We hypothesize that simulation-based training intervention will improve medical student competency in communicating bad news to patients.

ELIGIBILITY:
Inclusion Criteria:

* Residents working at the Intensive Care Unit.

Exclusion Criteria:

* Residents who are are available for the intervention or who don't have the appropriate number of meetings captured for data analysis

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-12 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with competency in communicating bad news behavioral measure | One month after training
  Number of Participants with competency in communicating bad news behavioral measure

CONTACTS AND LOCATIONS:
Overall Officials: Jingyuan Xu, M.D., Principal Investigator — Southeast University
Locations (1):
- Zhongda hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No